CLINICAL TRIAL: NCT00452972
Title: Complications of Exteriorized Versus In Situ Uterine Repair at Cesarean Delivery Under Spinal Anesthesia
Brief Title: Exteriorized Versus In Situ Uterine Repair at Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-04; 04-0057-A
Record Dates: First submitted 2007-03-19; First posted 2007-03-28 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: Vomiting; Nausea; Pain; Hypotension; Tachycardia
Keywords: Cesarean delivery; Spinal anesthesia; Nausea; Vomiting; Pain
MeSH Terms: conditions — Vomiting; Nausea; Pain; Hypotension; Tachycardia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Spinal Anesthesia

SUMMARY:
This study was undertaken to compare the two techniques (exteriorized vs in situ) of uterine repair with respect to patient comfort, hemodynamic changes, surgical time and blood loss, in patients undergoing elective CD under a strictly standardized spinal anesthetic. We hypothesized that in situ uterine repair would be more comfortable for the patients.

DETAILED DESCRIPTION:
Uterine repair during Cesarean delivery can be done either by exteriorizing the uterus and replacing it into the abdominal cavity after the completion of a double layer closure, or by suturing it in situ. Exteriorization of the uterus has been shown to decrease blood loss during Cesarean delivery when compared to in situ repair. However, at the same time, it is thought to be uncomfortable for the patient with respect to intraoperative nausea, vomiting and pain. Intraoperative nausea and vomiting in patients who receive regional anaesthesia for Cesarean section is a complex multifactorial problem arising from anesthetic and non-anesthetic causes. Additionally, it can influence hemodynamic stability.

The study was a prospective, randomized and single blinded study. It compared the effects of exteriorization of the uterus and in-situ repair during Cesarean delivery with respect to patient's comfort, hemodynamic changes, uterine contractility and blood loss in patients under spinal anesthesia. All low risk patients undergoing elective C-delivery under spinal anesthesia were considered for this study.

Spinal anesthesia was performed in the sitting position with 10-12 mg of 0.75% hyperbaric bupivacaine, mixed with 100 mcg of preservative free morphine and 10 mcg of fentanyl. Any drop in blood pressure was treated with 100 mg of phenylephrine titrated to maintain systolic blood pressure within 10% of the baseline values throughout the procedure. Oxytocin was used judiciously, in aliquots of 0.5 IU. Obstetricians were asked to allow assisted spontaneous delivery of placenta rather than manual extraction. During surgery, patient's complaints of nausea, vomiting, pain or any discomfort were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women scheduled for elective cesarean delivery

Exclusion Criteria:

* ASA III or IV patients
* Patient with conditions that predispose to uterine atony and post partum hemorrhage

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2004-04; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative nausea or vomiting after deliver of the infant

SECONDARY OUTCOMES:
Intraoperative pain
Calculated blood loss
Uterine contractility
Hypotension
Heart rate changes
Duration of uterine repair

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Siddiqui M, Goldszmidt E, Fallah S, Kingdom J, Windrim R, Carvalho JC. Complications of exteriorized compared with in situ uterine repair at cesarean delivery under spinal anesthesia: a randomized controlled trial. Obstet Gynecol. 2007 Sep;110(3):570-5. doi: 10.1097/01.AOG.0000277712.67230.22. PMID 17766602